CLINICAL TRIAL: NCT07214116
Title: Effectiveness of Educational Intervention, Virtual Reality, and Music Therapy on Anxiety in Onychocryptosis Surgery
Brief Title: Virtual Reality, Music, and Education to Reduce Anxiety in Patients Undergoing Ingrown Toenail Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Seville (Other)
Responsible Party: Principal Investigator, Raquel Prieto Domínguez, University Degree in Podiatry, University of Seville
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: SICEIA-2025-1206
Record Dates: First submitted 2025-10-02; First posted 2025-10-09 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Ingrown Toenail
Keywords: Ingrown toenail; Onychocryptosis; Virtual reality; Music therapy; Educational video; Podiatry; Pain management; preoperative anxiety
MeSH Terms: conditions — Nails, Ingrown; Agnosia | interventions — Music Therapy

STUDY DESIGN:
Intervention Model Description: Randomized, parallel assignment with three groups: (1) Control group receiving standard care without educational video, music, or virtual reality; (2) Experimental group 1 receiving an educational video combined with virtual reality; (3) Experimental group 2 receiving an educational video combined with music therapy. Groups will be compared to evaluate effectiveness in reducing anxiety and pain in onychocryptosis surgery.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (No Intervention): Participants undergo traditional onychocryptosis surgery without educational video, music, or virtual reality.
- Experimental group 1 (Experimental): Participants watch an educational video before the surgery and use virtual reality glasses during the onychocryptosis surgery.
  Interventions: Behavioral: Educational Video; Device: Virtual Reality
- Experimental group 2 (Experimental): Participants watch an educational video before the surgery and listen to music through headphones during the onychocryptosis surgery.
  Interventions: Behavioral: Educational Video; Behavioral: Music Therapy

INTERVENTIONS:
Behavioral: Educational Video — The educational video will last 5 minutes and is designed to inform participants about the onychocryptosis surgical procedure. The principal investigator will clearly and accessibly explain what the surgery involves, the steps to follow, and what participants can expect before, during, and after the procedure.
  Arms: Experimental group 1; Experimental group 2
Device: Virtual Reality — Participants will use Meta Quest 3 VR glasses during the onychocryptosis surgery. The device features adjustable straps, interpupillary distance settings, and built-in headphones with spatial sound, allowing immersive visualization and audio tailored to patient preferences. Disposable masks will be used for hygiene. The immersive content will be a 360-degree video of a relaxing walk through a forest accompanied by gentle music, starting 5 minutes before the procedure. Patients may remove the glasses or stop the VR experience at any time if desired.
  Other Names: VR; Virtual reality glasses; VR glasses; VR headset; Virtual reality headset
  Arms: Experimental group 1
Behavioral: Music Therapy — Participants will wear over-ear headphones with disposable covers and noise-cancellation (Bose® QuietComfort 25) connected to an Apple® iPod. Music will start 5 minutes before the ingrown toenail surgery and continue throughout the procedure. Only instrumental classical music, royalty-free and from Musopen.org, will be played in a 1-hour playlist. The same playlist will be used for all participants. Participants can adjust the volume at any time. Music will be temporarily paused if communication with the patient is needed and resumed afterward.
  Other Names: Music listening
  Arms: Experimental group 2

SUMMARY:
The main objective of this clinical trial is to evaluate whether watching an educational video before surgery, combined with the use of virtual reality or music during surgery, can reduce anxiety and pain in people undergoing ingrown toenail (onychocryptosis) surgery.

The main questions the study aims to answer are:

Are the educational video, virtual reality, and music effective in controlling and reducing pain and anxiety during surgery compared to traditional surgery?

As a distraction technique, is virtual reality or music more effective in reducing pain and anxiety during surgery?

Do these interventions produce changes in patients' physiological parameters during surgery?

Is there a relationship between patients' sociodemographic characteristics and their level of anxiety when undergoing surgery?

Three study groups will be compared to determine the effect of each intervention:

Experimental Group 1: watch a 5-minute educational video before entering the operating room and use virtual reality glasses with a 360° immersive video of a relaxing walk in the forest during surgery.

Experimental Group 2: watch the 5-minute educational video before surgery and listen to carefully selected instrumental music through noise-canceling headphones during surgery.

Control Group: surgery performed in the traditional way, without an educational video, virtual reality, or music.

All participants will complete questionnaires to assess anxiety, pain, and satisfaction before and after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older of any sex.
* Diagnosed with ingrown toenail (onychocryptosis) requiring surgical treatment.
* Cognitive ability to understand study information, follow instructions, and complete questionnaires.

Exclusion Criteria:

* Patients requiring ingrown toenail surgery associated with another pathology or surgical technique (e.g., subungual exostosis, chondroma, foreign bodies, tenotomies, etc.).
* Patients with difficulties understanding Spanish.
* Patients with visual or auditory disabilities preventing full use of the educational video, virtual reality, or headphones.
* Patients with a diagnosis of trait anxiety, depression, or any emotional disorder.
* Patients under psychiatric treatment.
* Patients with chronic foot pain.
* Patients receiving treatment for chronic pain.
* Patients with epilepsy.
* Patients with severe vertigo.
* Patients with current facial injuries or burns.
* Patients under treatment for blood pressure.
* Patients with coagulation disorders.
* Patients with active infections.
* Pregnant women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Generalized Anxiety Disorder Scale (GAD-7) | The scale will be completed by patients after viewing the educational video and before entering the operating room.
  The Generalized Anxiety Disorder Scale (GAD-7) is a brief questionnaire consisting of 7 questions designed to identify symptoms associated with generalized anxiety disorder. The questions refer to the last 15 days and are answered using a 4-point Likert scale (0 = not at all, 3 = nearly every day), with a maximum score of 21. Based on the final score, anxiety levels are classified into four categories: 0-4 (minimal), 5-9 (mild), 10-14 (moderate), and 15-21 (severe). In this study, the GAD-7 will be used to analyze the relationship between higher preoperative and intraoperative anxiety and the presence of generalized anxiety disorder.
The Amsterdam Preoperative Anxiety and Information Scale (APAIS) | The scale will be completed by patients after viewing the educational video and before entering the operating room.
  The Amsterdam Preoperative Anxiety and Information Scale (APAIS) is a self-administered 6-item questionnaire that evaluates preoperative anxiety and the patient's need for information regarding surgery. It consists of two subscales: APAIS-A (items 1, 2, 4, and 5), which measures anxiety with scores ranging from 4 (not anxious) to 20 (maximum anxiety), and APAIS-I (items 3 and 6), which measures the need for information and is classified into three levels: 2-4 (no additional information needed), 5-7 (moderate need), and 8-10 (high need). Each item is rated on a 5-point Likert scale, where 1 = "Not at all" and 5 = "Extremely," allowing to obtain clear information from surgical patients about both their level of anxiety and their need for information in the preoperative phase.
Preoperative Visual Analogue Scale for Anxiety (VAS-A pre) | Measured once after viewing the educational video and prior to entering the operating room.
  The Visual Analogue Scale for Anxiety (VAS-A) is a single-item tool used to assess anxiety. It consists of a 10 cm horizontal line anchored with the descriptors "not anxious at all" on the left end and "extremely anxious" on the right end. Patients are asked to place a mark on the line corresponding to their current level of anxiety. The score is obtained by measuring in millimeters from the left end of the line to the patient's mark, resulting in a range from 0 to 100, where higher values indicate greater anxiety. The VAS-A pre will be used to evaluate the patient's preoperative anxiety.
Intraoperative Visual Analogue Scale for Anxiety (VAS-A intra) | Measured once postoperatively, after the patient has left the operating room and is in the pre-recovery area.
  The Visual Analogue Scale for Anxiety (VAS-A) is a single-item tool used to assess anxiety. It consists of a 10 cm horizontal line anchored with the descriptors "not anxious at all" on the left end and "extremely anxious" on the right end. Patients are asked to place a mark on the line corresponding to their current level of anxiety. The score is obtained by measuring in millimeters from the left end of the line to the patient's mark, resulting in a range from 0 to 100, where higher values indicate greater anxiety. The VAS-A intra will be used to evaluate the patient's anxiety during the surgical procedure. To preserve the immersive experience in the operating room, this questionnaire will be completed after the surgery, but the scale clearly instructs the patient to report how they felt during the procedure
Postoperative Visual Analogue Scale for Anxiety (VAS-A post) | Measured once postoperatively, after the patient has left the operating room and is in the pre-recovery area.
  The Visual Analogue Scale for Anxiety (VAS-A) is a single-item tool used to assess anxiety. It consists of a 10 cm horizontal line anchored with the descriptors "not anxious at all" on the left end and "extremely anxious" on the right end. Patients are asked to place a mark on the line corresponding to their current level of anxiety. The score is obtained by measuring in millimeters from the left end of the line to the patient's mark, resulting in a range from 0 to 100, where higher values indicate greater anxiety. The VAS-A post will be used to evaluate the patient's anxiety after the surgical procedure.
State-Trait Anxiety Inventory - State-Anxiety Subscale (STAI-S) | Measured once postoperatively, after the patient has left the operating room and is in the pre-recovery area.
  The State-Anxiety subscale reflects a transient emotional condition, measuring the anxiety experienced at the present moment. It consists of 20 items, each rated on a 4-point Likert scale according to the intensity of perceived anxiety: 0 ("Almost never/Not at all"), 1 ("Somewhat/Sometimes"), 2 ("Moderately/Often"), and 3 ("Very much/Almost always"). Total scores range from 0 to 60. In this study, the STAI-State subscale will be used exclusively, as we aim to assess the anxiety experienced by the patient at the time of surgery. To preserve the immersive experience in the operating room, this questionnaire will be completed after the surgery, but the scale clearly instructs the patient to report how they felt during the procedure.
Visual Analogue Scale for Maximum Pain (VAS-P Max) | Measured once postoperatively, after the patient has left the operating room and is in the pre-recovery area.
  The Visual Analogue Scale for Pain (VAS-P) is a single-item tool used to assess pain intensity. It consists of a 10 cm horizontal line anchored with the descriptors "no pain" on the left end and "worst imaginable pain" on the right end. Patients are asked to place a mark on the line corresponding to their pain level. The score is obtained by measuring in millimeters from the left end of the line to the patient's mark, resulting in a range from 0 to 100, where higher values indicate greater pain. VAS-P Max will be used to record the highest level of pain experienced by the patient during surgery. To preserve the immersive experience in the operating room, this scale will be completed after the surgery, but the scale clearly instructs the patient to report how they felt during the procedure.
Visual Analogue Scale for Average Pain (VAS-P average) | Measured once postoperatively, after the patient has left the operating room and is in the pre-recovery area.
  The Visual Analogue Scale for Pain (VAS-P) is a single-item tool used to assess pain intensity. It consists of a 10 cm horizontal line anchored with the descriptors "no pain" on the left end and "worst imaginable pain" on the right end. Patients are asked to place a mark on the line corresponding to their pain level. The score is obtained by measuring in millimeters from the left end of the line to the patient's mark, resulting in a range from 0 to 100, where higher values indicate greater pain. VAS-P Average will be used to record the average pain experienced by the patient throughout the surgical procedure. To preserve the immersive experience in the operating room, this scale will be completed after the surgery, but the scale clearly instructs the patient to report how they felt during the procedure.

SECONDARY OUTCOMES:
Preoperative Systolic Blood Pressure | Measured once prior to the start of surgery, after 5 minutes of rest while the patient is seated.
  Systolic blood pressure will be measured in millimeters of mercury (mmHg) using a validated automatic blood pressure monitor, with the patient seated and after 5 minutes of rest. A single value will be recorded prior to the start of surgery to characterize the patient's baseline hemodynamic status.
Preoperative Diastolic Blood Pressure | Measured once prior to the start of surgery, after 5 minutes of rest while the patient is seated.
  Diastolic blood pressure will be measured in millimeters of mercury (mmHg) using a validated automatic blood pressure monitor, with the patient seated and after 5 minutes of rest. A single value will be recorded prior to the start of surgery to characterize the patient's baseline hemodynamic status.
Preoperative Heart Rate | Measured once prior to the start of surgery, after 5 minutes of rest while the patient is seated.
  Heart rate will be measured in beats per minute (bpm) using a validated automatic monitor or pulse oximeter, with the patient seated and after 5 minutes of rest. A single value will be recorded prior to the start of surgery to characterize the patient's baseline cardiovascular status.
Preoperative Oxygen Saturation | Measured once prior to the start of surgery, after 5 minutes of rest while the patient is seated.
  Oxygen saturation (SpO₂) will be measured as a percentage using a validated pulse oximeter, with the patient seated and after 5 minutes of rest. A single value will be recorded prior to the start of surgery to characterize the patient's baseline respiratory status.
Intraoperative Systolic Blood Pressure | Measured at four specific intraoperative moments: disinfection, anesthesia administration, first incision, and bandaging.
  Systolic blood pressure (mmHg) will be measured using a validated automatic blood pressure monitor at four predefined moments during the surgery: (1) disinfection of the surgical area, (2) application of local anesthesia, (3) first incision or invasive technique, and (4) final bandaging. This will allow monitoring of hemodynamic changes during the procedure.
Intraoperative Diastolic Blood Pressure | Measured at four specific intraoperative moments: disinfection, anesthesia administration, first incision, and bandaging.
  Diastolic blood pressure (mmHg) will be measured using a validated automatic blood pressure monitor at four predefined moments during the surgery: (1) disinfection of the surgical area, (2) application of local anesthesia, (3) first incision or invasive technique, and (4) final bandaging. This will allow monitoring of hemodynamic changes during the procedure.
Intraoperative Heart Rate | Measured at four specific intraoperative moments: disinfection, anesthesia administration, first incision, and bandaging.
  Heart rate (beats per minute) will be measured using a validated automatic monitor at four predefined moments during the surgery: (1) disinfection of the surgical area, (2) application of local anesthesia, (3) first incision or invasive technique, and (4) final bandaging. This will allow monitoring of cardiovascular response during the procedure.
Intraoperative Oxygen Saturation | Measured at four specific intraoperative moments: disinfection, anesthesia administration, first incision, and bandaging.
  Oxygen saturation (%) will be measured using a validated pulse oximeter at four predefined moments during the surgery: (1) disinfection of the surgical area, (2) application of local anesthesia, (3) first incision or invasive technique, and (4) final bandaging. This will allow monitoring of respiratory function during the procedure.
Postoperative Systolic Blood Pressure | Measured once postoperatively, after the patient has left the operating room and is in the pre-recovery area.
  Systolic blood pressure (mmHg) will be measured using a validated automatic blood pressure monitor once the patient has exited the operating room and is in the pre-recovery area. This measurement will assess the patient's hemodynamic status immediately after the surgery.
Postoperative Diastolic Blood Pressure | Measured once postoperatively, after the patient has left the operating room and is in the pre-recovery area.
  Diastolic blood pressure (mmHg) will be measured using a validated automatic blood pressure monitor once the patient has exited the operating room and is in the pre-recovery area. This measurement will assess the patient's hemodynamic status immediately after the surgery.
Postoperative Heart Rate | Measured once postoperatively, after the patient has left the operating room and is in the pre-recovery area.
  Heart rate (beats per minute) will be measured using a validated automatic monitor once the patient has exited the operating room and is in the pre-recovery area. This measurement will assess the patient's cardiovascular response immediately after the surgery.
Postoperative Oxygen Saturation | Measured once postoperatively, after the patient has left the operating room and is in the pre-recovery area.
  Oxygen saturation (%) will be measured using a validated pulse oximeter once the patient has exited the operating room and is in the pre-recovery area. This measurement will assess the patient's respiratory status immediately after the surgery.
Satisfaction with Received Information | Measured once, immediately before entering the operating room.
  Participants will rate their satisfaction with the information they have received regarding the surgical procedure using a 5-point Likert scale (1 = Not satisfied at all, 2 = Slightly satisfied, 3 = Neutral, 4 = Very satisfied, 5 = Completely satisfied). This measure will capture the patient's perception of the adequacy and clarity of preoperative information.
Satisfaction with Educational Video | Measured once, after reviewing the educational video and before entering the operating room.
  Participants in the experimental groups will rate their satisfaction with the educational video they have viewed prior to the surgery using a 5-point Likert scale (1 = Not satisfied at all, 2 = Slightly satisfied, 3 = Neutral, 4 = Very satisfied, 5 = Completely satisfied). This measure assesses the participant's perception of the video's usefulness and clarity. Participants in the control group will not complete this measure, as they will not have viewed the video.
Satisfaction with Surgical Procedure | Measured once postoperatively, after the patient has left the operating room and is in the pre-recovery area.
  Participants will rate their satisfaction with the surgical procedure they have just undergone using a 5-point Likert scale (1 = Not satisfied at all, 2 = Slightly satisfied, 3 = Neutral, 4 = Very satisfied, 5 = Completely satisfied). This measure captures the patient's perception of the quality and outcome of the surgery.
Satisfaction with Anesthesia | Measured once postoperatively, after the patient has left the operating room and is in the pre-recovery area.
  Participants will rate their satisfaction with the anesthesia administered during the surgical procedure using a 5-point Likert scale (1 = Not satisfied at all, 2 = Slightly satisfied, 3 = Neutral, 4 = Very satisfied, 5 = Completely satisfied). This measure captures the patient's perception of comfort and adequacy of anesthesia.
Satisfaction with Virtual Reality | Measured once postoperatively, after the patient has left the operating room and is in the pre-recovery area.
  Participants in the experimental group 1 will rate their satisfaction with the use of virtual reality glasses during the surgical procedure using a 5-point Likert scale (1 = Not satisfied at all, 2 = Slightly satisfied, 3 = Neutral, 4 = Very satisfied, 5 = Completely satisfied). This measure assesses the participant's experience and comfort with the virtual reality intervention. Participants in other groups will not complete this measure.
Satisfaction with Music Therapy | Measured once postoperatively, after the patient has left the operating room and is in the pre-recovery area.
  Participants in the experimental group 2 will rate their satisfaction with listening to music during the surgical procedure using a 5-point Likert scale (1 = Not satisfied at all, 2 = Slightly satisfied, 3 = Neutral, 4 = Very satisfied, 5 = Completely satisfied). This measure captures the participant's experience and comfort with the music intervention. Participants in other groups will not complete this measure.